CLINICAL TRIAL: NCT05280002
Title: Outcomes of Single Intra-articular Injection of Adipose-tissue-derived Total-Stromal-cells (TOST) Therapy in Knee Osteoarthritis
Brief Title: Adipose-tissue-derived Total-Stromal-cells (TOST) Therapy in Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Collaborators: Dhaka Medical College (Other)
Responsible Party: Principal Investigator, Moshiur Rahman Khasru, Associate Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSMMU/2018/25
Record Dates: First submitted 2022-02-24; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis Knees
Keywords: Osteoarthritis, Adipose Tissue, TOST, Stem Cell
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Both clinical and high-frequency-ultrasound-scanning Assessors were blinded about the case and control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adipose Tissue derived Total-Stromal-Cells (TOST) (Experimental): Adipose Tissue derived Total-Stromal-Cells (TOST) containing mesenchymal stem cells plus standard conservative care.
  Interventions: Biological: Adipose Tissue derived Total-Stromal-Cells (TOST)
- Control (No Intervention): Standard Conventional Treatment

INTERVENTIONS:
Biological: Adipose Tissue derived Total-Stromal-Cells (TOST) — Single dose autologous aAdipose Tissue derived Total-Stromal-Cells (TOST) containing mesenchymal stem cell was injected in each knee of the participants having knee osteoarthritis.
  Arms: Adipose Tissue derived Total-Stromal-Cells (TOST)

SUMMARY:
In this phase II Randomized Clinical Trial (RCT), impacts of a single Intra-articular injection of autologous adipose tissue derive total-stromal-cells (TOST) on knee pain, physical function, stiffness, and cartilage thickness assessed and compared changes before and after intervention.

Individuals with knee osteoarthritis (KOA) diagnosed by using the American College of Rheumatology (ACR) criteria for Osteoarthritis knee were included in the study. Kellgren-Lawrence (KL) radiological scores were used to define radiological changes and high-frequency musculoskeletal ultrasonogram (MSUS) was used to measure cartilage thickness.

DETAILED DESCRIPTION:
A phase II randomized clinical trial (RCT) was performed with primary Knee osteoarthritis (KOA) attended in the department of physical medicine and rehabilitation, BSMMU, between January 2018 and December 2021. Approval was obtained from the institutional review board of BSMMU for this clinical trial (Reference No: BSMMU/2018/25, dated 01/01/2018). Impacts of a single intra-articular (IA) injection of autologous adipose tissue derived total-stromal-cells (TOST) containing mesenchymal stem cells on pain, physical function, stiffness, and cartilage thickness assessed and compared before and after intervention. Patients satisfied the American College of Rheumatology (ACR) criteria for osteoarthritis (OA) knee included in the study. Kellgren-Lawrence (KL) radiological scores were used to define OA grade; however, high-frequency musculoskeletal ultrasonogram (MSUS) was used to measure cartilage thickness. There is no standard protocol to follow while assessing cartilage thickness; however, recent work of Podlipska and co-workers would be a worth consideration for using adipose tissue for cartilage regeneration. As medial tibio-femoral joint is the most commonly involved in KOA, here, we consider medial femoral cartilage thickness. The assessment used a commercially available ultrasound device (Samsung Accuvix, 2010, origin- South Korea) with a 15 megahertz linear transducer ML6-15. The patient was positioned supine with the knee in full flexion. A proximal-distal probe sweeping over the anterior-central knee area, medial femoral articular cartilage imaged in an axial plane. Degenerated cartilage signified either loss of surface sharpness or increased inner echogenicity; local or total thinning of articular cartilage. The definitions for articular cartilage degeneration are as follows: Grade 0 - a monotonous anechoic band with sharp hyperechoic anterior and posterior interfaces, Grade 1 - loss of the average sharpness of cartilage interfaces and or increased echogenicity of the cartilage, Grade 2a - grade 1 plus thinning of articular cartilage less than 50%, Grade 2b - more than 50% but less than 100% thinning of articular cartilage, Grade 3 -100% local loss of the cartilage tissue.

A total of thirty KOA was randomly divided into two groups - case and control. Both groups received conventional care for KOA (acetaminophen 1 gram thrice daily for 14 days, quadriceps strengthening exercises, aerobic exercise, mind-body, proprioception, mechanical diagnosis, and therapy (MDT) exercises, and activities of daily living (ADL) modifications4, 18-20. Fifteen received six milliliters (ml) single-dose of autologous adipose tissue derived total-stromal-cells (TOST) and 3 ml activated PRP). PRP was activated with 0.1 ml calcium gluconate per 0.9 ml of PRP (1:9 ratio). However, no orthobiological product was given in another fifteen participants.

ELIGIBILITY:
Inclusion Criteria:

* Primary KOA with KL-grade II and III radiological changes

Exclusion Criteria:

* KOA received IA steroid, viscosupplementation, or PRP injection or undergone knee surgery within the last six months.
* Patients with septic and tubercular arthritis, post-traumatic hemarthrosis, unstable knee joint due to anterior cruciate ligament (ACL) injury, malignancy, autoinflammatory arthritis (gout), inflammatory disease (rheumatoid arthritis, psoriatic arthritis, reactive, and ankylosing spondylitis), and charcot arthropathy.
* Patients with local eczematous skin and skin infection

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity | Before treatment and after treatment at week 4, 12, and 24
  Changes in pain intensity are assessed from baseline and at week 4, 12, and 24 using Visual Analogue scale (VAS) [0-10 cm scale], where score '0' denotes no pain and 10 means worst pain.
Changes in Physical functioning of knee joints. | Before treatment and after treatment at week 4, 12, and 24
  Changes in Physical functioning of knee joints were measured by The Western Ontario and McMaster Universities Arthritis Index (WOMAC). There are 17 items consist in WOMAC physical function such as Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties. Each item is scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The WOMAC physical score ranges between 0 and 68. The lower score means better knee functioning.
Changes in femoral cartilage thickness | Baseline and 24 weeks after treatment
  Changes in cartilage thickness was measured from baseline to 24 weeks of the study period using high frequency ultrasound 15 MHz (6-15 MHz) transducer (Samsung Accuvix, 2010, South Korea). Mean femoral cartilage was considered for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Moshiur Rahman Khasru, MBBS, FCPS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Decision is required from all the investigators on consensus basis.